CLINICAL TRIAL: NCT00285194
Title: hOKT3γ1 (Ala-Ala) Combined With Sirolimus and Delayed Tacrolimus in Type 1 Diabetic Islet Allograft Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0003M44181
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Type 1 Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — alanylalanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Allogeneic Islets of Langerhans
Drug: hOKT3γ1 (Ala-Ala)

SUMMARY:
The collective effects of two-layer pancreas preservation, pretransplant islet culture, day -2 pretransplant immunosuppression, and induction immunosuppression with the FcR-nonbinding anti-CD3 monoclonal antibody hOKT3γ1 (Ala-Ala)to facilitate diabetes reversal after single-donor islet transplantation.

DETAILED DESCRIPTION:
This is an open-label, one-year follow-up study of type 1 diabetic islet allograft recipients who receive FcR non-binding OKT3 antibody hOKT3γ1 (Ala-Ala) plus sirolimus induction immunotherapy combined with sirolimus and delayed tacrolimus maintenance immunosuppression. Six subjects were transplanted.

The premise behind the proposal is that hOKT3γ1(Ala-Ala) corrects the imbalance between autoreactive and regulatory T cells and consequently prevents autoimmune destruction of transplanted islets. To prevent allorejection, hOKT3γ1(Ala-Ala)was combined with sirolimus and delayed tacrolimus. Additionally, the safety and efficacy of the maintenance immunosuppressive regimen of sirolimus combined with tacrolimus was monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Primary islet allotransplant
2. Type 1 diabetes mellitus, complicated by at least one of the following situations that persist despite intensive efforts in close cooperation with their diabetes care team:

   1. Metabolic lability/instability;
   2. Reduced awareness of hypoglycemia;
   3. Persistently poor glucose control (as defined by HgbA1c>10% at the end of six months of intensive management efforts with the diabetes care team);
   4. Progressive secondary complications.
3. Age 18 and older
4. Able to give written informed consent

Exclusion Criteria:

1. Age less than 18 years
2. Body weight greater than75 kg.
3. BMI greater than 26 kg/m2 for male and females
4. Waist-to-hip ratio 0.80 (female) and 0.95 (male)
5. First degree relative with type 2 diabetes
6. Insulin requirement of greater than 0.7 IU/kg/day
7. HbA1C greater than 12%
8. Positive C-peptide response to intravenous arginine stimulation
9. Untreated proliferative retinopathy
10. Macroalbuminuria (urinary albumin excretion greater than 300 mg/24hrs)
11. Creatinine clearance greater than 85 ml/min/1.73 m2 in females, greater than 95 ml/min/1.73 m2 in males
12. Serum creatinine greater than 1.2 mg/dl
13. Previous pancreas or islet transplant
14. Previous OKT3 antibody therapy
15. Presence of history of panel-reactive anti-HLA antibodies greater than 10%
16. Abnormal T4 and TSH despite thyroid replacement therapy
17. Positive pregnancy test, or presently breast-feeding
18. Active infection
19. Negative screen for Epstein-Barr Virus (EBV) by an EBNA method
20. Invasive aspergillus infection within year prior to study entry
21. Any history of malignancy
22. Active alcohol or substance abuse
23. History of non-adherence to prescribed regimens
24. Psychiatric disorder making the subject not a suitable candidate for transplantation
25. Karnofsky performance score greater than 70
26. Baseline Hgb greater than 11.7 g/dl; lymphopenia (greater than 1,000/L), or leukopenia (greater than 4,000 total leukocytes/L), or an absolute CD4+ count <500/L
27. Thrombocytopenia greater than 150 x 109/L
28. Use of warfarin or other anticoagulant therapy (except aspirin) or patient with PT-INR greater than 1.5
29. Severe co-existing cardiac disease
30. Baseline liver function tests outside of normal range
31. Presence of gallstones on baseline ultrasound exam
32. Active peptic ulcer disease
33. Severe unremitting diarrhea or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications
34. Celiac disease
35. Hyperlipidemia (fasting LDL cholesterol greater than 130 mg/dl, treated or untreated; and/or fasting triglycerides greater than 200 mg/dl)
36. Addison's disease.
37. Under treatment for a medical condition requiring chronic use of systemic steroids
38. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2000-04; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, immune activity, and pharmacokinetics of hOKT3γ1 (Ala-Ala) antibody induction therapy for the prevention of autoimmune destruction and rejection of allogeneic islet transplants as measured by:
-Physical examination
-Vital signs
-Body weight
-Adverse events
-Laboratory and diagnostic safety assessments included complete blood counts with differential and platelets, circulating T cell phenotypes, and serum chemistry.
-Immune activity and pharmacokinetic assessments included hOKT3γ1 (Ala-Ala) level and half-life, monoclonal antibody coating and modulation of CD3 on peripheral blood T cells, and anti-hOKT3γ1 (Ala-Ala) antibody responses.

SECONDARY OUTCOMES:
Efficacy of hOKT3γ1 (Ala-Ala) antibody induction therapy for the prevention of autoimmune destruction and rejection of islet transplants as defined by:
-Proportion of subjects with full islet graft function (insulin independence and HbA1c <7%);
-Proportion of subjects with partial islet graft function (insulin dependence, basal or arginine-stimulated C-peptide levels of greater or equal to 0.5 ng/ml and HbA1c <7%);
-Proportion of subjects with slet graft loss will be defined as a return to insulin therapy for >30 days, absence of basal and arginine-stimulated C-peptide, re-transplantation, or patient death;

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard J. Hering, M.D., Principal Investigator — University of Minnesota
Locations (1):
- Universtiy of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Hering BJ, Kandaswamy R, Harmon JV, Ansite JD, Clemmings SM, Sakai T, Paraskevas S, Eckman PM, Sageshima J, Nakano M, Sawada T, Matsumoto I, Zhang HJ, Sutherland DE, Bluestone JA. Transplantation of cultured islets from two-layer preserved pancreases in type 1 diabetes with anti-CD3 antibody. Am J Transplant. 2004 Mar;4(3):390-401. doi: 10.1046/j.1600-6143.2003.00351.x. PMID 14961992
- See also: Diabetes Institute for Immunology and Transplantation - U of M — http://www.diabetesinstitute.org